CLINICAL TRIAL: NCT05846464
Title: Virtual Reality to Enhance Upper Extremity Physical Therapy and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Johns Hopkins University (Other); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: WRNMMC-2021-0376
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Injuries to the Hand and Wrist
Keywords: virtual reality; hand; therapy; immersive; take-home

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Virtual Reality to Enhance Upper Extremity Physical Therapy and Recovery (Experimental): This is a descriptive study assessing the feasibility of using VR rehabilitation with unilateral (or bilateral) impairment of the arm, wrist, and or hand resulting in reduced range of motion, dexterity, and/or strength of the hand. Phase I: Typical Home Exercise Program, Phase II: Use of VR headset in conjunction with current Home Exercise Program. Intervention sessions include the baseline, midpoint and final visits.
  Interventions: Device: Meta Quest 2

INTERVENTIONS:
Device: Meta Quest 2 — The Meta/Oculus Quest (along with the SignWave software) delivers an immersive audio/visual-based game environment where the users hand is created and displayed in the virtual environment and matches target gestures to the beat of the music.

SUMMARY:
This is a descriptive study assessing the feasibility of using VR rehabilitation with unilateral (or bilateral) impairment of the arm, wrist and or hand resulting in reduced range of motion, dexterity, and/or strength of the hand.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of using a virtual reality program to monitor and encourage compliance with musculoskeletal home exercise programs. It hypothesizes that the treatment will display improved compliance, range of motion, and general function for individuals with upper extremity musculoskeletal deficits.

The primary objectives are to: 1. Describe participant compliance with an immersive game-based virtual reality (VR) rehabilitation device for delivering at-home occupational therapy exercises for the wrist and hand in individuals with motor impairments. 2. Describe and compare functional outcomes among participants before and after completing at-home rehabilitation using the VR system.

These objective outcomes will be measured through various standardized tests completed by qualified study team members.

ELIGIBILITY:
Inclusion Criteria:

* DoD Beneficiary
* Exhibiting musculoskeletal impairment requiring continued at-home rehabilitation
* Cleared by research or clinical medical provider for participation
* Participant no longer has active range of motion movement restrictions. They may still have weight bearing restrictions but nothing that will preclude them from moving their hand and digits to their maximum ability.
* Ability to keep hand and arm in the field of view of the VR scene
* Must have demonstrated the ability for the Oculus to track all hand and wrist motions of interest (during an initial screening at baseline)
* Ability to independently don and doff the VR headset, plus start the app (verified in the Occupational Therapy/Physical Therapy clinic)
* Age range between 18-65
* Demonstrate the ability to tolerate wearing the VR headset

Exclusion Criteria:

* History of photo-induced seizures
* History of motion sickness when using VR equipment (especially vestibular effects such as nausea, dizziness, etc.)
* Partial amputations of the arm being assessed (including missing digits as they may not enable tracking by the VR)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Jebsen-Taylor Hand Function Test | 30 minutes
  Assessment of functional use and selection of appropriate grasp for common activities of daily living

SECONDARY OUTCOMES:
9-hole Peg Test | 10 minutes
  Speed and accuracy of grasp and release
Hand/wrist goniometric range of motion (ROM) | 15 minutes
  Hand/wrist range of motion assessment

OTHER OUTCOMES:
Quick DASH (Disabilities of the Arm, Shoulder and Hand) Questionnaire | 5 minutes
  Self-reported perception of functional ability of arm, shoulder, and hand
NASA-TLX | 5 minutes
  Ease of use preference and mental load survey
System Usability Scale | 2 minutes
  Quantitative ease of use assessment
Open-Ended Usability Scale | 2 minutes
  Qualitative ease of use assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No